CLINICAL TRIAL: NCT00864292
Title: Predictors of Neuro-cognitive Decline and Survival in HIV-infected Subjects
Status: Completed | Type: Observational
Sponsor: SEARCH Research Foundation (Other)
Collaborators: Thai Red Cross AIDS Research Centre (Other)
Responsible Party: Victor Valcour, John A. Burns School of Medicine, Honolulu, Hawaii
Other Study IDs: SEARCH 001.1
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2009-03

CONDITIONS: AIDS; Dementia
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV-infected, no dementia: Patients with HIV-infection but no dementia
- HIV-infected, dementia: Patients with HIV-infection and dementia

SUMMARY:
Patients will be followed every 6 months for a total of 5 visits (Month 0, 6, 12, 18 and 24). The first visit is the screening and entry visit which can occur at any time after the subject finishes SEARCH 001 study but preferably it should occur approximately 6 months after SEARCH 001 study completion.

At each visit, patients will undergo the following

1. Assessment of function including activity of daily living questionnaire
2. History of medical illnesses, medication history
3. Neurological examination: All patients will have a neurological evaluation and neuropsychological evaluation to characterize neurocognitive and neurological status. (It is possible that patients within the non-dementia group will meet criteria for dementia after close testing is completed).
4. Neuropsychological assessment:
5. Thai Depression Inventory.
6. HIV viral load and storage of blood for proviral DNA level

Final outcome assessment based on all available data. If possible, it is intended that these diagnoses will be determined through monthly VTC conference calls with UH investigators. This consensus conference will include the Thai investigators, the UH neurologist, the UH neuropsychologist and the UH principal investigators.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have completed the SEARCH 001 study are eligible to enroll in this SEARCH 001.1 study provided that they understand and voluntarily sign the informed consent form.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jintanat Ananworanich, PhD, Principal Investigator — SEARCH Research Foundation
Locations (1):
- South East Asia Research Collaboration with Hawaii, Bangkok, Thailand